CLINICAL TRIAL: NCT03000933
Title: Human Papillomavirus (HPV) Infection in Young Men Who Have Sex With Men Following Introduction of Universal Male HPV Vaccination Program in Australia
Brief Title: Human Papillomavirus in Young People Epidemiological Research 2 (HYPER2)
Acronym: HYPER2
Status: Completed | Type: Observational
Sponsor: The Alfred (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Eric Chow, Senior Research Fellow, The Alfred
Other Study IDs: Merck-54860
Record Dates: First submitted 2016-12-19; First posted 2016-12-22 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Human Papillomavirus; Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Oral sampling for HPV
  2. Anal sampling for HPV&
  3. Penile sampling for HPV
  4. Blood for HPV, HIV, Syphilis
  5. Anal swabs for rectal gonorrhoea and chlamydia
  6. Pharyngeal swabs for gonorrhoea and chlamydia
  7. Urine sample for gonorrhoea and chlamydia
  Oral, penile, and anal specimens will be collected from each man at two visits 7 days apart. Routine HIV and STI (chlamydia, gonorrhoea, and syphilis) screening will be performed at baseline (Day 0).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young same-sex attracted men: Same-sex attracted men aged 16 to 20

SUMMARY:
Australia was one of the countries to implement a universal school-based male vaccination program - in 2013. This research project will examine the prevalence of HPV among young men who have sex with men (MSM) who have been offered school-based HPV vaccination.

DETAILED DESCRIPTION:
HYPER-2, will be a cross-section study, using the same recruitment and testing strategies used in HYPER 1, which determined the prevalence of anal, genital and oral HPV among men who have sex with men aged 16-20 years. Given the differing age groups that will have been offered vaccination over the 2 study period, men aged 16-19 will be recruited in the first year (2017) and men aged 16-20 will be recruited in the second year (2018) to ensure that the participants included in the HYPER-2 study would have been eligible for the free male HPV vaccine in Australia. A total of 200 men will be recruited over a 2-year period, and HPV vaccination status for each participant will be verified against the National HPV Vaccination Program Register.

This 2-year cross-sectional study will recruit men who report sex with men aged from 16 to 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 16 to 20 (Must be aged 16-19 years from 1 January 2017 to 31 December 2017, and aged 16-20 years from 1 January 2018 to 31 December 2018)
* Report any previous type of sexual contact (including but not restricted to oral or anal sex) with at least one other man ever
* Able to complete all study requirements including questionnaire in English and completion of 2 visits
* Residing in Australia since 2013 (This is to ensure that males included in the study were present in Australia at the time HPV vaccination was offered)

Exclusion Criteria:

* Transgender male

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young same sex attracted men 16-20 years of age in Melbourne, Australia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of quadrivalent vaccine HPV types | Baseline
  The primary outcome of interest will be the prevalence of quadrivalent vaccine types (6, 11, 16 and 18) among 16-20 year old MSM and comparison of these with non-quadrivalent vaccine HPV types which would be expected to remain high unless there is significant cross protection. Oral, penile, and anal HPV prevalence will be calculated.

SECONDARY OUTCOMES:
Persistent HPV infection | Day 7
  Detection of same HPV type at the same site at both visits (day 0 and 7). The objective of repeat sampling at day 7 is to investigate whether this might distinguish transient HPV detection from infection. A brief questionnaire will be self-completed by participants at day 7 to ascertain whether there has been any sexual re-exposure between day 0 and 7 that might explain repeat HPV positivity at day 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Melbourne Sexual Health Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chow EPF, Tabrizi SN, Fairley CK, Wigan R, Machalek DA, Garland SM, Cornall AM, Atchison S, Hocking JS, Bradshaw CS, Balgovind P, Murray GL, Chen MY. Prevalence of human papillomavirus in young men who have sex with men after the implementation of gender-neutral HPV vaccination: a repeated cross-sectional study. Lancet Infect Dis. 2021 Oct;21(10):1448-1457. doi: 10.1016/S1473-3099(20)30687-3. Epub 2021 May 24. PMID 34043963
- [Result] Chow EPF, Fairley CK, Zou H, Wigan R, Garland SM, Cornall AM, Atchison S, Tabrizi SN, Chen MY. Human Papillomavirus Antibody Levels Following Vaccination or Natural Infection Among Young Men Who Have Sex With Men. Clin Infect Dis. 2022 Aug 25;75(2):323-329. doi: 10.1093/cid/ciab1052. PMID 34971362